CLINICAL TRIAL: NCT04158492
Title: Impact of Comprehensive Molecular Tests on Antimicrobial Stewardship in Community-acquired Pneumonia: an Open, Controlled and Randomized Clinical Trial
Brief Title: Impact of Comprehensive Molecular Tests on Antimicrobial Stewardship in Community-acquired Pneumonia
Acronym: RADICAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Fundació La Marató de TV3 (Other); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Jordi Carratala, Head of Infectious Diseases, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-INF-RADICAP
Record Dates: First submitted 2019-10-28; First posted 2019-11-08 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Community-acquired Pneumonia
Keywords: antimicrobial stewardship; point-of-care test; comprehensive molecular tests; multiple PCR
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Controlled, open-label clinical trial with two parallel groups (1:1) settled in two tertiary care hospitals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard diagnostic tests (Active Comparator): Patients who will undergo only the standard diagnostic procedures
  Interventions: Diagnostic Test: Standard diagnostic procedures
- Experimental + standard diagnostic tests (Experimental): Patients will undergo described standard diagnostic procedures and in addition, real-time multiplex Protein Chain Reaction (PCR, FilmArray Pneumonia panel Plus ™, Biofire, BioMérieux).
  Interventions: Diagnostic Test: real-time multiplex PCR

INTERVENTIONS:
Diagnostic Test: real-time multiplex PCR — Patients will be randomly assigned to receive experimental diagnosis (comprehensive molecular testing added to routine microbiological testing) AND standard diagnosis microbiological procedures
  Arms: Experimental + standard diagnostic tests
Diagnostic Test: Standard diagnostic procedures — Patients who will undergo only the standard microbiological diagnostic procedures: blood cultures, Gram stain and culture sputum when possible, Gram and pleural fluid culture when appropriate, urine determination of the pneumococcal and Legionella pneumophila serogroup antigens type 1. A serological study will be carried out for the etiological agents of atypical pneumonia in the acute and convalescent phases of the infection.
  Arms: Standard diagnostic tests

SUMMARY:
Background: Community-acquired pneumonia (CAP) continues to be a major health problem with significant mortality and it's one of the main causes of antibiotic prescription. Antibiotic overuse is a key driver of antimicrobial resistance and exposes patients to an increased risk of other antibiotic-related adverse events. The investigators aim to assess if rapid molecular tests are an effective tool to reduce antibiotic use in CAP compared to routine microbiological testing.

Design: Randomized, controlled, open-label clinical trial with two parallel groups (1:1) settled in a two-year multicenter, two tertiary care hospitals, between 2019 and 2021. Eligible participants will be non-severely immunosuppressed adult patients hospitalized for CAP through the emergency department. Primary endpoint will be antibiotic consumption measured by days of antibiotic therapy (DOT) per 1000 patient-days. Secondary end points will be: de-escalation to narrower antibiotic treatment, time to switch from intravenous to oral antibiotics, antibiotic-related side effects, length of hospital stay, days until clinical stability, need for ICU admission, need for hospital readmission in the 30 days after randomization, death from any cause in the 30 days after randomization. Patients will be randomly assigned to receive experimental diagnosis (comprehensive molecular testing added to routine microbiological testing) or standard diagnosis (only microbiological routine testing). A total of 220 patients are estimated in the experimental arm (undergoing comprehensive molecular testing) and 220 control subjects (undergoing routine testing) to be able to reject the null hypothesis that experimental and control groups have equal DOT per 1000 patients-days with a probability above 0.8.

Discussion: Comprehensive molecular tests could be a key tool in the optimization of etiological diagnostics in CAP and, therefore, a key element in antimicrobial stewardship programs developed to improve safety and antibiotic use in CAP.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older), of both sexes, hospitalized with a diagnosis of CAP in the first 24 hours of the admission.
* Patient or his legal representative gives the informed consent

Exclusion Criteria:

* Patient with acute infection by SARS-CoV-2 being this defined as:

  * Clinic of COVID-19 compatible, PCR positive for SARS-CoV-2 and negative serology for SARS-CoV-2.

OR

* COVID-19 clinic compatible, PCR positive for SARS-CoV-2 (in the last 60 days) and positive serology for SARS-CoV-2.

  * Pregnancy and / or nursing.
  * Severe immunocompromised patients (chemotherapy or radiotherapy in the previous 90 days, use of immunosuppressive drugs, chronic use of corticosteroids at a minimum dose of 15 mg / day in the last two weeks, transplantation of hematopoietic progenitors, solid organ transplant, patients with HIV and CD4 count ≤ 200 cells / mm3).
  * Imminent death (life expectancy ≤ 24 hours).
  * Participation in another clinical trial of pharmacological treatment during the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Number of DOT | Up to 30±5 days after hospital discharge
  Number of days of antibiotic therapy

SECONDARY OUTCOMES:
Number of days with intravenous antibiotic treatment. | Up to 30±5 days after hospital discharge
  Number of days of intravenous antibiotic treatment
Number of days until de-escalation | Up to 30±5 days after hospital discharge
  Number of days until de-escalation of antibiotic treatment to another of narrower spectrum
Number of days until antimicrobial monotherapy | Up to 30±5 days after hospital discharge
  Number of days untilt antimicrobial monotherapy
Number of days until etiological diagnosis | Up to 30±5 days after hospital discharge
  Number of days until detection of the causal agent
Number of days of Oxygen treatment | Up to 30±5 days after hospital discharge
  Days of oxygen treatment
Number of days of non-invasive ventilation | Up to 30±5 days after hospital discharge
  Days of invasive or non-invasive mechanical ventilation
Number of days of hospital admission | Up to hospital discharge - a medium of 5 days
  Number of days of hospital admission
Rate of readmissions | Up to 30±5 days after hospital discharge
  Rate of patients who are readmitted after hospital discharge
Rate of complicated community-acquired pneumonia (CAP) | Up to 30±5 days after hospital discharge
  Rate of complications related to CAP
Rate of general complications | Up to 30±5 days after hospital discharge
  Patients with medical complications not directly related to CAP until the end of the clinical trial.
Number of adverse events | Up to 30±5 days after hospital discharge
  Number of total adverse events.
Number of adverse events related to antimicrobials | Up to 30±5 days after hospital discharge
  Number of adverse events related to antibiotic therapy.
Number of participants with Clostridium difficile infection | Up to 30±5 days after hospital discharge
  Number of patients diagnosed with Clostridium difficile infection during the clinical trial.
Phlebitis rate | Up to 30±5 days after hospital discharge
  Number of patients with phlebitis resulting from the use of intravenous drugs.
Early mortality rate | Up tp 5 days after randomization
  Number of patients deceased 5 days after the randomization
30 day case-fatality rate | Up to 30±5 days after randomization
  Number of patients deceased 30±5 days after randomization
CAP-related fatality rate | Up to 30±5 days after hospital discharge
  Number of patients Deceased patients, related to CAP during the clinical trial
All-cause fatality rate | Up to 30±5 days after hospital discharge
  Number of patients who died from any cause during the clinical trial
Number of DOT per 1000 patients-day | Up to 30±5 days after hospital discharge
  Number of Days of antibiotic treatment per 1000 patients-day

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Carratalà Fernández, PhD, Study Director — Institut d'Investigació Biomèdica de Bellvitge
Locations (4):
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Moisés Broggi University Hospital, Sant Joan Despí, Barcelona
  - SCIAS Hospital de Barcelona, Barcelona, Catalonia
  - Hospital de Bellvitge, Barcelona

IPD SHARING:
Plan to Share IPD: No
Data will be made available after evaluating individual request.

REFERENCES:
- [Derived] Abelenda-Alonso G, Calatayud L, Rombauts A, Meije Y, Oriol I, Sopena N, Padulles A, Niubo J, Duarte A, Llaberia J, Aranda J, Gudiol C, Satorra P, Tebe C, Ardanuy C, Carratala J. Multiplex real-time PCR in non-invasive respiratory samples to reduce antibiotic use in community-acquired pneumonia: a randomised trial. Nat Commun. 2024 Aug 17;15(1):7098. doi: 10.1038/s41467-024-51547-8. PMID 39154071
- [Derived] Kerneis S, Visseaux B, Armand-Lefevre L, Timsit JF. Molecular diagnostic methods for pneumonia: how can they be applied in practice? Curr Opin Infect Dis. 2021 Apr 1;34(2):118-125. doi: 10.1097/QCO.0000000000000713. PMID 33395094
- [Derived] Abelenda-Alonso G, Rombauts A, Gudiol C, Meije Y, Clemente M, Ortega L, Ardanuy C, Niubo J, Padulles A, Videla S, Tebe C, Carratala J. Impact of comprehensive molecular testing to reduce antibiotic use in community-acquired pneumonia (RADICAP): a randomised, controlled, phase IV clinical trial protocol. BMJ Open. 2020 Aug 20;10(8):e038957. doi: 10.1136/bmjopen-2020-038957. PMID 32819999